CLINICAL TRIAL: NCT00700726
Title: Study of the Patterns of Microvesicles in the Serum of Participants With Atopic and Non-atopic Asthma
Brief Title: Cohort Study of the Patterns of Microvesicles in the Serum of Participants With Atopic and Non-atopic Asthma
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Mastronarde, MD, John Mastronarde M.D., Ohio State University
Other Study IDs: 2007H0102
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Asthma; Allergies
Keywords: blood test; asthma; skin test
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, nasal lavage (optional)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A.: participants with atopic and non-atopic asthma

SUMMARY:
The purpose of this study is to determine if a simple blood test can help in disease management, particularly asthma. This will be researched by looking at certain features of the blood and to compare asthmatics without allergies to those that have allergy-induced asthma.

DETAILED DESCRIPTION:
A total of 20 participants (men or women) between the ages of 18-50 years with asthma will be enrolled. Participants will remain on their usual asthma treatments as prescribed by their usual asthma care provider. Current asthma treatments and any changes will be recorded at baseline and each subsequent visit. The primary outcome measures are correlation of microvesicle patterns with atopic state and variation from baseline with episodes of poor asthma control. Secondary outcomes include correlations between microvesicle patterns and spirometry, eNO levels, and glucorcorticoid sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18 and 50.
* have diagnosed asthma.
* must have less "one pack per day for 10 years" smoking history

Exclusion Criteria:

* You have had a fever of 100.4º within 24 hours of Visit 2.
* You are enrolled in another interventional research trial.
* Have other major chronic illnesses that would interfere with participation in the study.
* You are pregnant.
* You chronically use oral corticosteroids.
* You have taken anti-coagulants, insulin, and any investigative drugs within 2 months.
* You have the inability or unwillingness to provide consent.
* Inability to perform aerobic exercise.
* Inability to perform baseline measurements.
* Less than 80% completion of screening period diaries.
* Inability to be contacted by telephone.
* Intention to move out of the area within 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
correlation of microvesicle patterns with atopic state and variation from baseline with episodes of poor asthma control | 6 months

SECONDARY OUTCOMES:
correlations between microvesicle patterns and spirometry, eNO levels, and glucorcorticoid sensitivity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clay M. Marsh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Univeristy Medical Center, Columbus, Ohio, United States